CLINICAL TRIAL: NCT02773810
Title: Can Integration of Family Planning Services Into Anticoagulation Monitoring Services Improve Uptake of Long-Acting Reversible Contraception?
Brief Title: Integration of Family Planning Services Into Anticoagulation Monitoring Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Caitlin Bernard, Volunteer Clinical Assistant Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1504431629
Record Dates: First submitted 2016-05-11; First posted 2016-05-16 (Estimated); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Integrated Family Planning Services (Experimental): Women who agree to enrollment will undergo our intervention, which will include an educational intervention and free on-site provision of all reversible contraceptive options, including LARC. This educational 5 intervention will be a one-on-one educational session on all available methods of contraception, with an emphasis on the safety and efficacy of long-acting reversible contraception (LARC) and the importance of planning a pregnancy in women with medical conditions requiring anticoagulation. A provider (clinic officer, nurse or physician) trained in family planning counseling and provision will provide all counseling and discussions in Kiswahili. Women will then be offered free, on-site provision of whichever contraceptive method they choose by a trained provider.
  Interventions: Other: Integrated Family Planning Services

INTERVENTIONS:
Other: Integrated Family Planning Services — Women who agree to enrollment will undergo our intervention, which will include an educational intervention and free on-site provision of all reversible contraceptive options, including LARC. This educational 5 intervention will be a one-on-one educational session on all available methods of contraception, with an emphasis on the safety and efficacy of long-acting reversible contraception (LARC) and the importance of planning a pregnancy in women with medical conditions requiring anticoagulation. A provider (clinic officer, nurse or physician) trained in family planning counseling and provision will provide all counseling and discussions in Kiswahili. Women will then be offered free, on-site provision of whichever contraceptive method they choose by a trained provider.

SUMMARY:
Currently there are approximately 400 women of reproductive age enrolled in outpatient monitoring of warfarin therapy through AMS. The investigators do not have any data on the percentage of women who are using family planning, but anecdotally the providers report that it is very low. The investigators believe that an educational intervention with an emphasis on the safest and most effective methods, long-acting reversible contraception (LARC), aimed specifically toward women with medical conditions requiring anticoagulation, combined with on-site provision of LARC can improve uptake of these methods. Ultimately, the use of the most effective methods of contraception will prevent unplanned pregnancy and the unnecessary maternal morbidity and mortality associated with high-risk pregnancies in women with these conditions.

DETAILED DESCRIPTION:
The investigators' hypothesis is that implementation of an educational intervention emphasizing long-acting reversible contraception (LARC) combined with free on-site provision of LARC within Anticoagulation Monitoring Service (AMS) can improve uptake of these methods by 250% in this population.

Our objectives are to:

1. Determine whether integration of education about and free provision of highly effective long-acting reversible contraceptive methods within Anticoagulation Monitoring Services (AMS) is feasible.
2. Determine whether integration of education about and free provision of highly effective long-acting reversible contraceptive methods within Anticoagulation Monitoring Services (AMS) can improve uptake of long-acting reversible contraceptive methods (IUCDs and contraceptive implants).
3. Determine whether integration of education about and free provision of highly effective long-acting reversible contraceptive methods within an Anticoagulation Monitoring Services (AMS) Clinic can prevent unplanned pregnancies.

The investigators will perform a prospective cohort study of all women of reproductive age seen in Anticoagulation Monitoring Service (AMS). Women who agree to enrollment will undergo our intervention, which will include an educational intervention and free on-site provision of all reversible contraceptive options, including LARC. This educational intervention will be a one-on-one educational session on all available methods of contraception, with an emphasis on the safety and efficacy of long-acting reversible contraception (LARC) and the importance of planning a pregnancy in women with medical conditions requiring anticoagulation. A provider (clinic officer, nurse or physician) trained in family planning counseling and provision will provide all counseling and discussions in Kiswahili. Women will then be offered free, on-site provision of whichever contraceptive method they choose by a trained provider. During the intervention period we intend to capture all women currently actively enrolled in AMS, which is currently approximately 400 women. Each woman generally attends AMS clinic once per month, so the investigators expect that it will take about three months to capture all women at least once. These women will then be followed prospectively over the next one-year time period to evaluate for uptake of a contraceptive method and subsequent pregnancy. The investigators will then compare participants' method of contraception used prior to the intervention and participants' method of contraception used after the intervention. The investigators will specifically evaluate for an increase in the use of IUCDs and contraceptive implants.

ELIGIBILITY:
Inclusion Criteria:

* All women of reproductive age (age 14 to 50 or menopause) actively enrolled in Anticoagulation Monitoring Service (AMS) during the study timeframe.

Exclusion Criteria:

* Women who are pregnant.
* Women who have had a hysterectomy.
* Women who do not speak Kiswahili.

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 218 (Actual)
Dates: Start 2014-04; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Percent of women who have initiated the use of contraception | 3 months Post-intervention
  Proportion of women who initiated contraception after study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Bernard, MD, Principal Investigator — Indiana University

IPD SHARING:
Plan to Share IPD: No